CLINICAL TRIAL: NCT06275971
Title: Effectiveness of Continuous Glucose Monitoring System Among Cardiac Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, MD. PhD, Kangbuk Samsung Hospital, Sungkyunkwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2022-07-006
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Disease; PreDiabetes; Diabetes Mellitus
Keywords: continuous glucose monitoring
MeSH Terms: conditions — Heart Diseases; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Treatment group: glycemic control using CGM Control group: glycemic control using arterial/venous blood sampling and POCT glucose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CGM arm (Experimental): Glycemic control was monitored using CGM data for seven days following cardiac surgery
  Interventions: Device: Dexcom G6
- SMBG or venous/arterial glucose arm (Active Comparator): Glycemic control was monitored using SMBG or venous/arterial glucose data for seven days following cardiac surgery
  Interventions: Device: SMBG or venous/arterial blood glucose

INTERVENTIONS:
Device: Dexcom G6 — Glycemic control was monitored using CGM data for seven days following cardiac surgery
  Arms: CGM arm
Device: SMBG or venous/arterial blood glucose — Glycemic control was monitored using SMBG or venous/arterial blood glucose data for seven days following cardiac surgery
  Arms: SMBG or venous/arterial glucose arm

SUMMARY:
The aim of this study is to assess the level of glycemic control and the incidence of surgery-related complications in cardiac patients post-surgery when Continuous Glucose Monitoring (CGM) is utilized, as compared to traditional methods of arterial/venous blood sampling and Point-of-Care Testing (POCT) for glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subjects waiting for Elective Cardiac Surgery (CABG, Cardiac Valve Operation, Congenital heart anomaly surgery, aortic surgery, etc.)
* Subjects over the age of 18
* Patients with type 2 diabetes
* Patients with prediabetes

  1. HbA1c 5.7% or more
  2. fasting blood glucose 100 mg/dL or more
  3. 2 hours 75g-OGTT 140 mg/dL or more

Exclusion Criteria:

* Emergency surgery patients
* Patients performing co-operation other than cardiac surgery
* Patients with type 1 diabetes
* Total Pancreatectomy patients
* Patients with high surgical severity (STS score of 8 or more or EURO score of 5 or more)
* Patients who do not consent to the study
* Severe patients who are deemed difficult to continue research during surgery (excluded at the researcher's discretion)

  1. Cases where severe weight gain and severe edema occur after surgery
  2. Cases where the surgery time is significantly longer than average
  3. Cases where cardiopulmonary bypass is used more than once during surgery
* Others who are deemed unsuitable for research progression at the researcher's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Time within the target range of 100-180 mg/dL | 1-7 days after surgery
  Time within the target range of 100-180 mg/dL as assessed by CGM for 7 days after surgery

SECONDARY OUTCOMES:
Time within the target range of 100-140 mg/dL | 1-7 days after surgery
  Time within the target range of 100-140 mg/dL as assessed by CGM for 7 days after surgery
Time within the target range of 70-180 mg/dL | 1-7 days after surgery
  Time within the target range of 70-180 mg/dL as assessed by CGM for 7 days after surgery
Time to reach <70 mg/dL | 1-7 days after surgery
  Time to reach <70 mg/dL as assessed by CGM for 7 days after surgery
Time to reach <54 mg/dL | 1-7 days after surgery
  Time to reach <54 mg/dL as assessed by CGM for 7 days after surgery
Time to reach >180 mg/dL | 1-7 days after surgery
  Time to reach >180 mg/dL as assessed by CGM for 7 days after surgery
Time to reach >250 mg/dL | 1-7 days after surgery
  Time to reach >250 mg/dL as assessed by CGM for 7 days after surgery
Standard Deviation (SD) | 1-7 days after surgery
  SD value evaluated by CGM for 7 days after surgery
Coefficient of variation (CV) | 1-7 days after surgery
  CV value evaluated by CGM for 7 days after surgery
Mean glucose | 1-7 days after surgery
  Mean glucose value evaluated by CGM for 7 days after surgery
Glucose management indicator (GMI) | 1-7 days after surgery
  GMI value evaluated by CGM for 7 days after surgery
Number of days of ICU hospitalization | From 1 day after surgery until the date of ICU discharge or date of death from any cause, whichever came first, asessed up to 30 days
  Number of days of ICU hospitalization
Number of days hospitalized after surgery | From 1 day after surgery until the date of hospital discharge or date of death from any cause, whichever came first, asessed up to 30 days
  Number of days hospitalized after surgery
Number of participants with pneumonia occurrence after surgery | 1-7 days after surgery
  Number of participants with pneumonia occurrence within 1 week after surgery
Number of participants with wound infection occurrence after surgery | 1-7 days after surgery
  Number of participants with wound infection occurrence within 1 week after surgery
Number of participants who underwent CRRT implementation after surgery | 1-7 days after surgery
  Number of participants who underwent CRRT implementation within 1 week after surgery
Number of participants with Atrial fibrillation occurrence after surgery | 1-7 days after surgery
  Number of participants with Atrial fibrillation occurrence within 1 week after surgery
Number of participants with symptomatic CVA (ischemic and hemorrhagic) occurrence after surgery | 1-7 days after surgery
  Number of participants with symptomatic CVA (ischemic and hemorrhagic) occurrence within 1 week after surgery
Changes in concentration of serum CRP level after surgery | 1-7 days after surgery
  Changes in concentration of serum CRP level after surgery (between baseline and peak value within 1 week after surgery)
Mortality within 30 days of surgery | 1-30 days after surgery
  Mortality within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sun Joon Moon, MD, Study Director — Kangbuk Samsung Hospital, Sungkyunkwan University
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon SJ, Kim MS, Kim YT, Lee HE, Lee YW, Lee SJ, Chung ES, Park CY. Use of an insulin titration protocol based on continuous glucose monitoring in postoperative cardiac surgery patients with type 2 diabetes and prediabetes: a randomized controlled trial. Cardiovasc Diabetol. 2025 May 14;24(1):210. doi: 10.1186/s12933-025-02747-z. PMID 40369552